CLINICAL TRIAL: NCT00552747
Title: The Effect of Fenofibrate on Endothelial Function and HDL in Patients With Coronary Heart Disease and LDL-C at Goal
Brief Title: Effect of Fenofibrate on Endothelial Function and High-density Lipoproteins (HDL)in Patients With Coronary Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart Institute, Mexico (Other Government)
Responsible Party: Carlos Posadas-Romero MD, National Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fenofibrate
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Heart Disease; Hyperlipidemia
Keywords: fenofibrate; coronary heart disease; mixed hyperlipidemia
MeSH Terms: conditions — Coronary Disease; Hyperlipidemias; Hyperlipoproteinemia Type II | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): fenofibrate 160 mg capsules (QD) Taken once daily with the largest meal of the day
  Interventions: Drug: fenofibrate
- 2 (Placebo Comparator): placebo (capsules identical to those of fenofibrate) taken once daily (QD)with the largest meal of the day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fenofibrate — fenofibrate 160 mg capsules qd
  Arms: 1
Drug: placebo — capsules placebo
  Arms: 2

SUMMARY:
Fenofibrate is a drug that acts on the PPAR alpha receptors, increasing HDL-cholesterol and decreasing triglyceride levels. The interaction with these receptors has antiatherogenic actions by regulating the expression con key proteins that participate in vascular inflammation, plaque stability and thrombosis.

Fenofibrate reduces triglycerides and increases HDL-C in plasma. It also decreases small, dense LDL particles. The use of this drug has resulted in improvement of vascular function measured by endothelial function. Our hypotheses state that fenofibrate will improve: endothelial function, improve HDL antioxidant capacity and size distribution towards a predominance of small HDL particles.

DETAILED DESCRIPTION:
Patients with stable coronary heart disease, with LDL-C levels at goal will be invited to participate in this randomized, double blind study to receive either placebo or fenofibrate in addition to their statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18-60 years of age
* Stable coronary heart disease (no cardiovascular event 3 months prior to enrollment)
* Stable lipid-modifying drug therapy (previous 2 months)
* Low-dose statin therapy with LDL-C at goal (< 100 mg/dl)
* Triglyceride levels 151-500 mg/dl
* HDL-C levels <40 mg/dl

Exclusion Criteria:

* Diabetes mellitus
* Uncontrolled hypertension Systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg
* Subjects with renal (serum creatinine >1.5 times the upper limit of normal (ULN)), hepatobiliary (cholelithiasis, biliary cirrhosis, AST and/or ALT >2x ULN) or active thyroid disease (TSH >1.5x ULN or <0.05 uUI/ml)
* Hypersensitivity to fenofibrate or to any other component of its formula
* History of photoallergic reaction or phototoxicity to fenofibrate or ketoprofen

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
endothelial function | 8 weeks

SECONDARY OUTCOMES:
HDL particle distribution | 8 weeks
HDL associated antioxidant capacity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Posadas-Romero, MD, Principal Investigator — Principal Investigator; Pedro Reyes, MD, Study Director — head bioethics committee
Locations (1):
- Endocrinology Department National Institute of Cardiology Ignacio Chavez, Mexico City, Mexico

REFERENCES:
- [Background] Randomised trial of cholesterol lowering in 4444 patients with coronary heart disease: the Scandinavian Simvastatin Survival Study (4S). Lancet. 1994 Nov 19;344(8934):1383-9. PMID 7968073
- [Background] Shepherd J, Cobbe SM, Ford I, Isles CG, Lorimer AR, MacFarlane PW, McKillop JH, Packard CJ. Prevention of coronary heart disease with pravastatin in men with hypercholesterolemia. West of Scotland Coronary Prevention Study Group. N Engl J Med. 1995 Nov 16;333(20):1301-7. doi: 10.1056/NEJM199511163332001. PMID 7566020
- [Background] Sacks FM, Pfeffer MA, Moye LA, Rouleau JL, Rutherford JD, Cole TG, Brown L, Warnica JW, Arnold JM, Wun CC, Davis BR, Braunwald E. The effect of pravastatin on coronary events after myocardial infarction in patients with average cholesterol levels. Cholesterol and Recurrent Events Trial investigators. N Engl J Med. 1996 Oct 3;335(14):1001-9. doi: 10.1056/NEJM199610033351401. PMID 8801446
- [Background] Downs JR, Clearfield M, Weis S, Whitney E, Shapiro DR, Beere PA, Langendorfer A, Stein EA, Kruyer W, Gotto AM Jr. Primary prevention of acute coronary events with lovastatin in men and women with average cholesterol levels: results of AFCAPS/TexCAPS. Air Force/Texas Coronary Atherosclerosis Prevention Study. JAMA. 1998 May 27;279(20):1615-22. doi: 10.1001/jama.279.20.1615. PMID 9613910
- [Background] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Background] LaRosa JC, Grundy SM, Waters DD, Shear C, Barter P, Fruchart JC, Gotto AM, Greten H, Kastelein JJ, Shepherd J, Wenger NK; Treating to New Targets (TNT) Investigators. Intensive lipid lowering with atorvastatin in patients with stable coronary disease. N Engl J Med. 2005 Apr 7;352(14):1425-35. doi: 10.1056/NEJMoa050461. Epub 2005 Mar 8. PMID 15755765
- [Background] Gordon DJ, Probstfield JL, Garrison RJ, Neaton JD, Castelli WP, Knoke JD, Jacobs DR Jr, Bangdiwala S, Tyroler HA. High-density lipoprotein cholesterol and cardiovascular disease. Four prospective American studies. Circulation. 1989 Jan;79(1):8-15. doi: 10.1161/01.cir.79.1.8. PMID 2642759
- [Background] Hokanson JE, Austin MA. Plasma triglyceride level is a risk factor for cardiovascular disease independent of high-density lipoprotein cholesterol level: a meta-analysis of population-based prospective studies. J Cardiovasc Risk. 1996 Apr;3(2):213-9. PMID 8836866
- See also: National Institute of Cardiology Mexico City MEXICO — http://www.cardiologia.org.mx